CLINICAL TRIAL: NCT01776086
Title: Neuropsychological Testing Using Mobile Devices
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no subjects agreed to participate
Sponsor: Englewood Hospital and Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: E-12-471
Record Dates: First submitted 2013-01-23; First posted 2013-01-25 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Inpatients With Normal Neurological Function
MeSH Terms: interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Normal patients (Other): for patients with normal score on neurological testing with Folstein Mini-Mental Status Exam will then take the Scenes Task
  Interventions: Behavioral: Neurological testing

INTERVENTIONS:
Behavioral: Neurological testing
  Other Names: Scenes Task; Folstein Mini-Mental Status Exam

SUMMARY:
The purpose of this studying is to develop and characterize neuropsychological testing software for evaluating the prefrontal and temporal function of patients. As no software has been used for this purpose, this study will gather pilot data on the baseline performance of patients in a hospital setting that lack any neurological impairment. After creating this baseline, later experiments can be proposed to compare the performance in normal subjects with those who have neurologic injury or disease.

ELIGIBILITY:
Inclusion Criteria:

* Inpatients > = 18 years of age
* Patient must be able to provide informed consent

Exclusion Criteria:

* Patients with score of < 26 on Folstein Mini-Mental Status Exam
* Patients with known brain lesions
* Patients with history of stroke, neurologic disease or dementia
* Patients with acute illness or who are in imminent distress

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Determination of "normal performance" curve | 1 year
  The purpose of this study is to generate a curve of "normal performance" on the neurological test for hospitalized patients of different ages

CONTACTS AND LOCATIONS:
Overall Officials: James Young, MD, PhD, Principal Investigator — Englewood Hospital and Medical Center
Locations (1):
- Englewood Hospital and Medical Center, Englewood, New Jersey, United States